CLINICAL TRIAL: NCT04804202
Title: Virtual Cycling Environments (VCYCLE) Increases Exercise Intensity of Persons With Parkinson Disease
Brief Title: Virtual Cycling Environments for Persons With Parkinson Disease
Acronym: VCYCLE_PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Aging (NIA) (NIH); New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Judith E Deutsch, PT, PhD, Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro202000518; R15AG063348-01 (NIH)
Record Dates: First submitted 2021-03-02; First posted 2021-03-18 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
Keywords: virtual reality; exercise; cardiovascular intensity; neuromuscular intensity; enjoyment
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Repeated Measures Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual Reality (Other): This is a single arm study in which all participants will execute the same tasks over two sessions.
  Interventions: Other: Bicycling with and without virtual reality

INTERVENTIONS:
Other: Bicycling with and without virtual reality — In one session: Exercise intensity and enjoyment are measured while participants bicycle in a virtual compared to non-virtual environment. Cycling takes places in two modes continous and interval. In a second session exercise intensity and enjoyment are compared during bicycling with virtual reality presented in two different ways.

SUMMARY:
This study asks three questions about Persons with Parkinson Disease that use a bicycle for exercise. 1. Does the use of virtual reality increase the intensity and and enjoyment of the experience compared to bicycling without virtual reality? 2. Does the way in which the bicycling (interval compared to continous) is performed affect the experience? 3. How does the way the virtual reality is delivered (with goggles or projected on a screen) affect the experience?

DETAILED DESCRIPTION:
Participants attend two sessions. They complete movement assessments and questionnaires about physical activity. During the first session they bicycle in a semi-immersive (projected on a screen) and an immersive (with googles) virtual environment. After each bout they completed a questionnaire about the experience. In the second session they bicycle four times with and without a virtual environment using both a continous and interval mode. Their oxygen consumption is measured during cycling. They complete questionnaires after each exercise bout.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's disease
2. Hoehn and Yahr stages II-III,
3. 45-75 years old
4. able to ride a stationary upright bicycle
5. able to sign informed consent.

Exclusion Criteria:

1. Have a recent history of severe heart disease, severe lung disease, uncontrolled diabetes, traumatic brain injury or neurological disorder other than Parkinson Disease.
2. Are unable to follow directions or sign a consent form
3. Do not have adequate vision or hearing ability to see or hear a television
4. Have unstable medical condition or musculoskeletal disorder such as severe arthritis, recent knee surgery, hip surgery, or any other condition that the investigators determine would impair the ability to ride the bicycle
5. Have any other medical condition that prevents bicycling
6. Have moderate depression

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular Intensity | Collected in two sessions: Session 1(day 1 for 2 hours) collected continuously during 2 exercise bouts to compare exercise bouts.____Session 2 (day 2 for 2 hours) collected continuously in four exercise bouts to compare exercise bouts
  bicycling cadence collected continuously
Physiological Responses to Exercise- Oxygen Consumption | Collected in two sessions: Session 1(day 1 for 2 hours) collected continuously during 2 exercise bouts to compare exercise bouts___ Session 2 (day 2 for 2 hours) collected continuously in four exercise bouts to compare exercise bouts
  Metabolic equivalents derived from oxygen consumption which is collected continuously during four exercise bouts.
Enjoyment-Motivation | Collected in two sessions: Session 1 collected continuously during 2 exercise bouts in a 2 hour Session 2: in four exercise bouts in a 2 hour session to compare exercise bouts
  Intrinsic Motivation Inventory Enjoyment sub-scales collected at the end of each exercise bout
Heart Rate % of maximum | Collected in two sessions: Session 1 collected continuously during 2 exercise bouts in a 2 hour Session 2: in four exercise bouts in a 2 hour session to compare exercise bouts
  Collected continuously during exercise bouts and will be evaluated as a % of age adjusted maximum heart rate

SECONDARY OUTCOMES:
Borg Scale for Rate of perceived exertion | Collected in both Day 1 and 2 (each day is two hours) as follows: Day 1 (4 times in each of the two cycling bouts) Day 2 (6 times each of the four cycling bouts)
  Self-Report of Effort collected at a multiple time points to compare with exercise bouts
Cyber sickness Questionnaire | Collected in Day 1 (2 hour session) twice to compare before and after scores
  16 item questionnaire about feelings or symptoms of cyber sickness
Perceived Effort Ranking | Collected in once in day 1 and once in day 2
  Rating of Bicycling Conditions relative to each other (and audio recording of experience)
Enjoyment Ranking | Collected in once in day 1 and once in day 2
  Rating of Bicycling Conditions relative to each other (and audio recording of experience)

OTHER OUTCOMES:
UPDRS-III Subscale | Collected once in Day 1
  Description of Motor Performance Scored from 0-108 a lower score is better outcome
Physical Activity Scale for the Elderly | Collected once in Day 1
  Exercise Inventory Questionnaire
Geriatric Depression Scale (short form) | Collected once during Day 0 (screening)
  15 item inventory to rate depression (scored from 0-15 with a lower score being better)

CONTACTS AND LOCATIONS:
Overall Officials: Judith E. Deutsch, PT PhD, Principal Investigator — Rutgers
Locations (2):
- United States (2):
  - School of Health Professions, Newark, New Jersey
  - New York Institute of Technology, Old Westbury, New York

IPD SHARING:
Plan to Share IPD: Yes
Immediately following completion of our proposed study we will submit a de-identified data set of our protocol and links to published papers.
Supporting Information: Study Protocol
Time Frame: We will make study data available immediately following completion.
Access Criteria: Open Access